CLINICAL TRIAL: NCT07278375
Title: Target Trial Emulation for Pharmacologic Treatment of Neonatal Opioid Withdrawal Syndrome
Acronym: TreaT NOW
Status: Not yet recruiting | Type: Observational
Sponsor: HELP for NOWS Consortium (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: HELP for NOWS 03; 1U24HD107621 (NIH); 1UG1HD107628 (NIH); 1UG1HD107580 (NIH); 1UG1HD107649 (NIH); 1UG1HD107650 (NIH); 1UG1HD107653 (NIH); 1UG1HD107627 (NIH); 1UG1HD107631 (NIH); 1UG1HD107616 (NIH)
Record Dates: First submitted 2025-11-21; First posted 2025-12-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Opioid Withdrawal Syndrome
Keywords: Neonatal Opioid Withdrawal Syndrome; NOWS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants treated with buprenorphine: Infants treated with buprenorphine as the primary opioid for NOWS
- Infants treated with morphine: Infants treated with morphine as the primary opioid for NOWS

SUMMARY:
The goal of this observational study is to learn how two medicines used in routine care-buprenorphine and morphine-affect recovery in newborns (≥36 weeks' gestation) with Neonatal Opioid Withdrawal Syndrome (NOWS). The main questions it aims to answer are:

1. Do infants treated with buprenorphine become medically ready for discharge sooner than those treated with morphine?
2. Does one treatment lead to better overall clinical outcomes than the other?

Researchers will compare infants who received buprenorphine with infants who received morphine to see whether one treatment helps babies recover more quickly.

Participants will not be asked to do anything. Instead, the study team will collect information already documented in the infant's and mother's medical records securely without any contact or changes to clinical care.

No new medicines, procedures, or visits are involved. This study only reviews existing clinical data to better understand which commonly used treatment may support faster recovery for newborns with NOWS.

DETAILED DESCRIPTION:
Neonatal Opioid Withdrawal Syndrome (NOWS) occurs in infants who were exposed to opioids during pregnancy and may lead to symptoms such as irritability, feeding difficulties, and trouble sleeping. Many hospitals treat these symptoms with either morphine or buprenorphine, but it is not yet known whether one medication helps infants recover more quickly. This study aims to answer that question by reviewing information already documented in medical records from hospitals that routinely use one of these treatments.

The study will include approximately 796 infants, all born at 36 weeks' of gestation or later and treated for NOWS with either buprenorphine or morphine as part of usual clinical care. Data will be collected from about 22 hospitals across the United States. Researchers will review existing medical record information such as the infant's birth characteristics, withdrawal symptoms, details of treatment (including medication choice and dosing approach), feeding practices, non-pharmacologic care, and clinical outcomes-including the key measure of how long it took for the infant to become medically ready for discharge.

Because treatment decisions are made by the clinical team and not assigned by the study, researchers will use advanced statistical methods to compare outcomes between infants who received buprenorphine and those who received morphine. These methods allow the team to adjust for differences between infants and hospitals, helping ensure that comparisons are as fair and accurate as possible. The goal is to estimate how outcomes would differ if all infants received one medication versus the other in real-world practice.

No infants or parents will be contacted for this study, and no additional treatments, tests, or procedures will be performed. All data come from routine clinical care. The regulatory review for this project determined that informed consent from families is not required because the study uses only existing medical information and does not involve any interaction with participants or changes to medical care. All collected data will be handled securely and in compliance with federal privacy requirements.

The information learned from this research may help improve care for future infants with NOWS by providing clearer evidence on how commonly used treatments compare in supporting recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Infant is ≥ 36 weeks' gestational age
2. Infant had antenatal opioid exposure identified by at least one of the following:

   1. History of maternal opioid use during the second and/or third trimester of pregnancy as noted in the mother's or infant's medical record;
   2. Positive maternal toxicology screen for opioids during the second or third trimester of pregnancy; and/or
   3. Positive infant toxicology screen for opioids during the initial hospital stay.
3. The infant is being assessed and managed for NOWS at an eligible study site.
4. The infant is at risk for pharmacologic treatment for NOWS defined by either of the following:

   * At least 1 score ≥ 8 if assessed and managed with the Finnegan Neonatal Abstinence Scoring Tool (FNAST) or modification thereof
   * At least 1 "yes" if assessed and managed with the Eat, Sleep, Console (ESC) care approach
5. Infant met all inclusion criteria on or after March 25, 2024.

Exclusion Criteria:

1. Infant has major congenital anomalies.
2. Infant has neonatal encephalopathy (inclusive of hypoxic ischemic encephalopathy), a metabolic disorder, stroke, intracranial hemorrhage, or meningitis diagnosed prior to the initiation of pharmacologic treatment.
3. Infant is receiving respiratory support (any positive pressure or oxygen therapy) at 48 hours of age.
4. Infant has undergone major surgical intervention prior to or at 48 hours of age.
5. Infant has postnatal opioid exposure prior to the initiation of pharmacologic treatment for NOWS.
6. Infant was outborn and pharmacologic treatment was initiated at the transferring hospital.

Min Age: 0 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include infant and mother dyads who fulfill the study inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 796 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Time from birth until infant meets criteria for medically ready for discharge (count) | From date of birth until date of infant meeting criteria for medically ready for discharge (estimated to be < 90 days).
  Number of days from birth until infant meets criteria for medically ready for discharge. An infant is considered medically ready for discharge when they are discharged by the medical provider or when they meet both of the following criteria:
  * 96 hours of age
  * 48 hours since last dose of treatment with morphine or buprenorphine

SECONDARY OUTCOMES:
Length of hospital stay (count) | From date of birth until date of hospital discharge (estimated to be < 90 days).
  Number of days between birth and hospital discharge
Length of primary opioid treatment (count) | From date of birth until date of last primary opioid dose administration (estimated to be < 90 days).
  Number of days between the first and the last primary opioid dose administered
Number of primary opioid doses administered (count) | From date of birth until date of last primary opioid dose administration (estimated to be < 90 days).
  Number of primary opioid doses administered (count)
Receipt of secondary medication (binary) | From date of birth until date of first non-opioid secondary medication administration or until date of hospital discharge, whichever comes first (estimated to be < 90 days).
  Receipt of at least one dose of any amount of phenobarbital, clonidine, or some other non-opioid medication as a secondary medication
Inpatient composite safety outcome (binary) | From date of birth until date of first occurrence of seizure or excessive weight loss more than 15% from birthweight or until date of last primary opioid dose administration, whichever comes first (estimated to be < 90 days).
  Occurrence of at least one of the following events between birth and the last primary opioid dose administered:
  * Seizures
  * Excessive weight loss more than 15% from birthweight
Inpatient composite critical safety outcome (binary) | From date of birth until date of first occurrence of non-accidental trauma or death or until date of last primary opioid dose administration, whichever comes first (estimated to be < 90 days).
  Occurrence of at least one of the following events between birth and the last primary opioid dose administered:
  * Non-accidental trauma
  * Death
Inpatient composite safety outcome after receipt of pharmacologic treatment (binary) | From date of first primary opioid dose administration until date of first occurrence of seizure or excessive weight loss more than 15% from birthweight or until date of hospital discharge, whichever comes first (estimated to be < 90 days).
  Occurrence of at least one of the following events between first primary opioid dose administered and the data of hospital discharge:
  * Seizures
  * Excessive weight loss more than 15% from birthweight
Inpatient composite critical safety outcome after receipt of pharmacologic treatment (binary) | From date of first primary opioid dose administration until date of first occurrence of non-accidental trauma or death or until date of hospital discharge, whichever comes first (estimated to be < 90 days).
  Occurrence of at least one of the following events between first primary opioid dose administered and hospital discharge:
  * Non-accidental trauma
  * Death

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - ChristianaCare, Wilmington, Delaware
  - University of South Florida Health, Tampa, Florida
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana
  - University of Louisville Hospital, Jeffersonville, Indiana
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Children's Regional Hospital, Cooper University Health Care, Camden, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University of Rochester Medical Center, Rochester, New York
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Utah Health, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored at the DCC, RTI International. NIH Helping to End Addiction Long-term Initiative (HEAL) and NICHD requirements for data-sharing will apply. NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. In accordance with these policies (available at HEAL Public Access and Data Sharing | NIH HEAL Initiative), we will share de-identified data collected for the study. After the study is completed, the de-identified, archived data will be transmitted to a NIH HEAL supported repository, for use by other researchers including those outside of the study.
Supporting Information: Study Protocol, SAP
Time Frame: Within 1 year of study completion.

REFERENCES:
- See also: Study Portal — https://helpfornows.rti.org/